CLINICAL TRIAL: NCT00176527
Title: A Phase II Trial of 13-Cis Retinoic Acid, Alpha Interferon, Taxotere, and Estramustine (R.I.T.E.) for the Treatment of Hormone Refractory Prostate Cancer
Brief Title: Isotretinoin, Interferon Alfa-2b, Docetaxel, and Estramustine in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual goal met
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert DiPaola, MD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540176; P30CA072720 (NIH); CINJ#080107-3850
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Introns; Docetaxel; Estramustine; Isotretinoin; Electrophoresis, Polyacrylamide Gel; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: recombinant interferon alfa-2b
Drug: docetaxel
Drug: estramustine phosphate sodium
Drug: isotretinoin
Genetic: polyacrylamide gel electrophoresis
Genetic: protein expression analysis
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Isotretinoin may help prostate cancer cells become more like normal cells, and to grow and spread more slowly. Interferon alfa-2b may interfere with the growth of tumor cells. Drugs used in chemotherapy, such as docetaxel and estramustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving isotretinoin and interferon alfa-2b together with docetaxel and estramustine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving isotretinoin and interferon alfa-2b together with docetaxel and estramustine works in treating patients with metastatic prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate, in terms of change in measurable disease or prostate-specific antigen levels, in patients with hormone-refractory metastatic prostate cancer treated with isotretinoin, recombinant interferon alfa-2b, docetaxel, and estramustine phosphate sodium.

Secondary

* Determine the effect of this regimen on bcl-2 family proteins in peripheral blood mononuclear cell samples obtained from these patients.

OUTLINE: Patients receive oral isotretinoin once daily on days 1-4, recombinant interferon alfa-2b subcutaneously once daily on days 1-4, oral estramustine phosphate sodium three times daily on days 1-5, and docetaxel IV over 1 hour on day 2. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Peripheral blood mononuclear cells are acquired via blood draw at baseline and on days 2, 3, or 4 and analyzed for bcl-2 protein by IHC and electrophoresis.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hormone-refractory metastatic prostate cancer

  * Patients who have been recently withdrawn from treatment with bicalutamide or flutamide must demonstrate progression of disease
* Measurable disease OR prostate-specific antigen level ≥ 10 ng/mL

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Estimated life expectancy ≥ 6 months
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 8 g/dL
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* Bilirubin normal
* AST, ALT, and alkaline phosphatase (AP) must meet 1 of the following criteria:

  * AP normal and AST and ALT ≤ 2.5 times upper limit of normal (ULN)
  * AP elevated and AST and ALT normal
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No peripheral neuropathy > grade 1
* No concurrent active infections
* No concurrent major depression or suicidal ideation
* No concurrent medical condition that would preclude study participation
* No known HIV positivity
* Fertile patients must use effective contraception during and for 10 weeks after completion of study therapy

PRIOR CONCURRENT THERAPY:

* Recovered from prior surgery or radiotherapy
* No prior chemotherapy, retinoids, or interferon therapy
* More than 4 weeks since prior flutamide
* More than 6 weeks since prior bicalutamide

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2002-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response (biochemical and measurable disease)
Bcl-2 modulation in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. DiPaola, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States